CLINICAL TRIAL: NCT06737237
Title: Cervical Plexus Versus Infiltration for Clavicular Operations (CERPICO)
Acronym: CERPICO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Naval Medical Center Camp Lejeune (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Lee, Principal Investigator, Naval Medical Center Camp Lejeune
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCCL.2024.0027; NMCCL.2024.0027 (Other: NMCCL)
Record Dates: First submitted 2024-12-06; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Clavicle Surgery; Clavicle Fracture; Acromioclavicular Joint; Coracoclavicular Ligament
Keywords: clavicle surgery; cervical plexus block; local infiltration analgesia
MeSH Terms: interventions — Cervical Plexus Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Clinical Research Coordinator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided cervical plexus block (Active Comparator): u/s guided cervical plexus block will be performed with active local anesthetic, while the surgeon-administered local infiltration analgesia will be performed with placebo (0.9% sodium chloride)
  Interventions: Procedure: cervical plexus block; Procedure: Local Infiltration Analgesia (LIA)
- local infiltration analgesia (Active Comparator): surgeon-administered local infiltration analgesia will be performed with active local anesthetic, while the u/s guided cervical plexus block will be performed with placebo (0.9% sodium chloride)
  Interventions: Procedure: Local Infiltration Analgesia (LIA); Procedure: cervical plexus block

INTERVENTIONS:
Procedure: cervical plexus block — local anesthetic (10ml of bupivacaine 5mg/ml)
  Arms: ultrasound guided cervical plexus block
Procedure: Local Infiltration Analgesia (LIA) — local anesthetic (20ml of bupivacaine 2.5mg/ml)
  Arms: local infiltration analgesia
Procedure: cervical plexus block — placebo (10ml of 0.9% sodium chloride)
  Arms: local infiltration analgesia
Procedure: Local Infiltration Analgesia (LIA) — placebo (20ml of 0.9% sodium chloride)
  Arms: ultrasound guided cervical plexus block

SUMMARY:
Clavicle fractures are the most common fracture of the shoulder girdle, with young men being the most affected demographic. The incidence of clavicle fracture among military service members is 1.5-3x higher than the general adult population. While many clavicle fractures may be managed non-operatively, surgical intervention for clavicular fractures has shown improved functional outcomes in the active-duty Marine Corps population and an overall satisfactory return-to-duty rate. However, surgical fixation of the clavicle is associated with significant postoperative pain when no local anesthetic techniques are employed.

Several regional anesthetic and local infiltrative analgesic regimens have been studied to improve postoperative pain control for clavicle ORIF with the authors concluding that intermediate cervical plexus block is the regional anesthesia therapy of choice for post-operative analgesia. A retrospective study by the same group determined that an intermediate cervical plexus block resulted in lower postoperative pain scores and opioid requirements than surgeon-administered local infiltration analgesia. This retrospective study unfortunately lacked participant blinding, randomization, a standardized anesthetic, consistent block technique, and protocolized postoperative analgesia. To date, no prospective trial has been performed directly comparing these two techniques. We propose, given the significance of clavicle fractures and corrective surgery in the military population, to study the efficacy of ultrasound-guided intermediate cervical plexus blocks as compared to local infiltration analgesia.

DETAILED DESCRIPTION:
ALL PATIENTS (STANDARD CARE)

Patients will be administered a standardized anesthetic plan of preoperative anxiolysis (midazolam 2mg) and induction of anesthesia (lidocaine 1-1.5mg/kg, fentanyl 0.5-1.5mcg/kg, propofol 1-3mg/kg, and rocuronium 0.6-1.2mg/kg). Airway management will be at the discretion of the staff anesthesia provider.

Following endotracheal intubation, the anesthesia provider will perform an ultrasound-guided intermediate cervical plexus block. Ultrasound imaging will be used to identify the sternocleidomastoid muscle at its midpoint between origin and insertion. An echogenic needle will be advanced under live ultrasound guidance just deep to the posterior aspect of the sternocleidomastoid muscle.

UGICPB ARM (RESEARCH PROCEDURE)

LIA ARM (RESEARCH PROCEDURE)

10ml of bupivacaine 5mg/ml will be injected in 2ml aliquots with intermittent aspiration under direct visualization to confirm appropriate solution propagation and to avoid intravascular injection.

10ml normal saline will be injected in 2ml aliquots with intermittent aspiration under direct visualization to confirm appropriate solution propagation and to avoid intravascular injection.

ALL PATIENTS (STANDARD CARE)

Patients will then be administered a standardized anesthetic maintenance plan consisting of sevoflurane to age-adjusted MAC of >0.5, acetaminophen 1000mg IV, dexamethasone 10mg IV, ketorolac 30mg IV, tranexamic acid 1000mg IV, and rocuronium for neuromuscular blockade as indicated. The antibiotic regimen will be at the discretion of the orthopedic surgeon. For intraoperative pain control, the anesthesia provider will administer fentanyl 25-100mcg q5 min for HR and/or BP >20% baseline attributable to pain in the judgment of the anesthesia provider. No alternative opioids or adjuncts, such as nitrous oxide, ketamine, or dexmedetomidine, will be administered.

UGICPB ARM (RESEARCH PROCEDURE)

LIA ARM (RESEARCH PROCEDURE)

Prior to wound closure, the orthopedic surgeon will infiltrate the anticipated surgical site with 20ml of normal saline using a landmark-based technique.

Prior to wound closure, the orthopedic surgeon will infiltrate the anticipated surgical site with 20ml of bupivacaine 2.5mg/ml using a landmark-based technique.

ALL PATIENTS (STANDARD CARE)

Intermittent aspiration will be performed to avoid intravascular injection. The injectate will be evenly distributed along the skin, subcutaneous plane, musculature, and periosteum.

All patients will receive sugammadex 2-4mg/kg for reversal of neuromuscular blockade prior to emergence. Ondansetron 4mg may be given at the discretion of the staff anesthesia provider. Airway management for extubation will be at the discretion of the staff anesthesia provider; however, patients will not be transported to the PACU until emerged from general anesthesia.

On arrival to the PACU, the PACU nurse will perform their normal duties, including recording the times of PACU admission and discharge, initial and maximum pain score during phase 1 recovery, pain score at time of discharge, presence of nausea, administration of anti-emetic medication, emetic events, and incidence of Horner's syndrome in the patient's chart.

The PACU nurse will also, as a part of their normal duties, administer fentanyl per the standard institutional order set (25mcg fentanyl every 5 minutes as needed for pain score 1-4, 50mcg fentanyl every 10 minutes as needed for pain score 5-6, and 50mcg fentanyl every 5 minutes as needed for pain score 7-10) in the event rescue analgesia is indicated, up to a maximum of 250 mcg while in recovery phase 1. If the subject's pain continues to be uncontrolled after the administration of 250 mcg of fentanyl, or if the risk of continued opioid administration outweighs the benefit (in the opinion of the PACU anesthesia provider), alternative analgesics may then be utilized at the discretion of said PACU anesthesia provider. Additionally, the PACU nurse will record

Patients will be discharged with 800mg ibuprofen every 8 hours as needed, 1000mg acetaminophen every 8 hours as needed, and 5mg oxycodone every 6 hours as needed (15 tablets) for post-discharge analgesia, as is standard.

ALL PATIENTS (RESEARCH PROCEDURE)

After the patient has been discharged from the PACU, the Primary Investigators will retroactively collect the data from the OR and PACU that has been recorded in the patient's chart by their treatment providers. Note that the Primary Investigators will not make any treatment decisions or patient assessments, only record the existing information that other healthcare providers have collected.

Before discharge, the patient will receive a one-page pain diary on which to record answers regarding their pain level for the first 24-36 hours, to aid them in recalling their pain details for the post-op phone call.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64 years
* Scheduled surgery of the clavicle, acromioclavicular joint, or coracoclavicular ligament at NMCL
* ASA Physical Status Classification 1-3

Exclusion Criteria:

* Emergent surgery
* Concurrent surgery involving the glenobumeral joint or proximal humerus
* Prior anaphylactic reaction or known intolerance to study medications
* Patient reported or documented opioid use within the last 30 days unrelated to clavicular, AC joint, or CC ligament pathology

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Total Perioperative Intravenous Fentanyl Administration | from anesthesia start time to discharge from PACU, estimated 3-4 hours
  total fentanyl dosage (mcg) encompassing the intraoperative and PACU recovery periods

SECONDARY OUTCOMES:
PACU Pain Scores | from time of PACU admission to time of PACU discharge, estimated 30-60 minutes
  PACU pain score on time of PACU admission (0-10 on Numeric Pain Rating Scale), maximum pain score during PACU (0-10 on Numeric Pain Rating Scale), and pain score on discharge from PACU (0-10 on Numeric Pain Rating Scale)
PACU Rescue Analgesia | from time of PACU admission to time of PACU discharge, estimated 30-60 minutes
  The need for non-fentanyl analgesic medications during PACU recovery (yes/no)
Post-discharge Pain Scores | Night-of-surgery to postoperative day one
  Lowest pain score (0-10 on Numeric Pain Rating Scale), highest pain score (0-10 on Numeric Pain Rating Scale), average pain score (0-10 on Numeric Pain Rating Scale)
Postdischarge Oral Narcotic Use | Night-of-surgery to postoperative day one
  Quantity of oxycodone 5mg oral tablets required from night-of-surgery to postoperative day one
Postdischarge rebound pain | Night-of-surgery to postoperative day one
  The difference between pain scores (0-10 on Numeric Pain Rating Scale) when local anesthetic effect began to wear off and when local anesthetic effect wore off completely
Return to Emergency Room Rate | Night-of-surgery to postoperative day one
  The need to return to the emergency room for pain control from night-of-surgery to postoperative day one (yes/no)
Patient Satisfaction with Analgesia | End-of-surgery to postoperative day one
  The patient's overall satisfaction with postoperative pain management (Likert five-point scale, 1 being very dissatisfied to 5 being very satisfied)
PACU Adverse Event Rate | from time of PACU admission to time of PACU discharge, estimated 30-60 minutes
  The rate of PACU nausea/vomiting (yes/no), respiratory depression (yes/no), motor block (yes/no), and horner's syndrome (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: CDR Lee, MD, Principal Investigator — DHA/MD365
Locations (1):
- Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT06737237/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT06737237/ICF_001.pdf